CLINICAL TRIAL: NCT06135194
Title: Efficacy and Safety of T-Dxd in the Treatment of HER2-positive Breast Cancer With Brain Metastases After Prior Pyrotinib Treatment
Brief Title: Efficacy of T-Dxd in the Treatment of HER2-positive BCBM After Prior Pyrotinib
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing 302 Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: DS8021-Brain metastases
Record Dates: First submitted 2023-11-13; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — trastuzumab deruxtecan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: T-DXd — Efficacy and safety of T-DXd in the treatment of HER2-positive breast cancer with brain metastases after treatment with pyrotinib
  Other Names: DS-8201

SUMMARY:
To evaluate the efficacy and safety of T-DXd in the treatment of HER2-positive breast cancer with brain metastases after treatment with pyrotinib

ELIGIBILITY:
Inclusion Criteria:

(1) Women ≥18 years of age :(2) pathological diagnosis of HER2-positive breast cancer, defined as positive immunohistochemistry detection (+++) or FISH(Fluorescent In Situ Hybridization); (3) Imaging evidence of brain metastases; (4) Progression of brain metastases after prior treatment with pyrotinib, defined as progression of new or pre-existing brain metastases during treatment with pyrotinib; (5)ECOG score ≤3 points; (6) The efficacy of T-DXd should be evaluated at least once after treatment; (7) Bone marrow and organ functions are basically normal; (8) Complete medical records

Exclusion Criteria:

* Has uncontrolled or significant cardiovascular disease
* Has history of (noninfectious) interstitial lung disease (ILD)/pneumonitis that required steroids, has current ILD/pneumonitis, or suspected ILD/ pneumonitis that cannot be ruled out by imaging at screening
* Has any medical history or condition that per protocol or in the opinion of the investigator is inappropriate for the study

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with brain metastases from HER2 positive breast cancer after treatment with pyrotinib
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Central neryous system Progression Free Survival，CNS-PFS | 3years
  The interval from the start of treatment to the onset of disease progression or death from any cause in the intracranial lesions

SECONDARY OUTCOMES:
Overall Response Rate (ORR)for intracranial and extracranial lesions | 3years
  Percentage of patients with CompleteResponse (CR) and partial response (PartialResponse (PR)
Overall Clinical Benefit Rate (CBR) for intracranial and extracranial lesions | 3years
  Percentage of patients with complete response, partial response, and StableDisease (SD)≥6 months
Overall survival (Oversall Survival, OS) and security | 5years
  The interval between the start of treatment and death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: tao wang, Study Director — Beijing 302 Hospital
Locations (1):
- The Fifth Medical Center of PLA General Hospital, Beijing, Beijing Municipality, China